CLINICAL TRIAL: NCT04182113
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) as a Probe of Episodic Memory (EM) Neurocircuitry in Schizophrenia
Brief Title: rTMS as a Probe of Episodic Memory Neurocircuitry in Schizophrenia
Acronym: rTMS-EM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tom Hummer, Assistant Research Professor of Psychiatry, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1907931487
Record Dates: First submitted 2019-10-28; First posted 2019-12-02 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; psychosis; early phase psychosis; rTMS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: All patients will receive 1 Hz rTMS, 20 Hz rTMS, and Sham rTMS, in a randomized order.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (6):
- 1 Hz rTMS Stimulation first, then 20 Hz rTMS Stimulation, then sham rTMS (Experimental): Subjects will receive one session of each: low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of motor threshold (MT), for a total of 1200 pulses, high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minute, Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
  Interventions: Device: 1 Hz rTMS Stimulation; Device: Sham rTMS Stimulation
- 1 Hz rTMS Stimulation first, then sham rTMS, then 20 Hz rTMS Stimulation (Experimental): Subjects will receive one session of each: low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of motor threshold (MT), for a total of 1200 pulses, high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minute, Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
  Interventions: Device: 1 Hz rTMS Stimulation; Device: Sham rTMS Stimulation
- 20 Hz rTMS Stimulation first, then 1 Hz rTMS Stimulation, then sham rTMS (Experimental): Subjects will receive one session of each: low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of motor threshold (MT), for a total of 1200 pulses, high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minute, Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
  Interventions: Device: 1 Hz rTMS Stimulation; Device: Sham rTMS Stimulation
- 20 Hz rTMS Stimulation first, then sham rTMS, then 1 Hz rTMS Stimulation (Experimental): Subjects will receive one session of each: low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of motor threshold (MT), for a total of 1200 pulses, high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minute, Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
  Interventions: Device: 1 Hz rTMS Stimulation; Device: Sham rTMS Stimulation
- sham rTMS first, then 1 Hz rTMS Stimulation, then 20 Hz rTMS Stimulation (Experimental): Subjects will receive one session of each: low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of motor threshold (MT), for a total of 1200 pulses, high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minute, Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
  Interventions: Device: 1 Hz rTMS Stimulation; Device: Sham rTMS Stimulation
- sham rTMS first, then 20 Hz rTMS Stimulation, then 1 Hz rTMS Stimulation (Experimental): Subjects will receive one session of each: low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of motor threshold (MT), for a total of 1200 pulses, high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minute, Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
  Interventions: Device: 1 Hz rTMS Stimulation; Device: Sham rTMS Stimulation

INTERVENTIONS:
Device: 1 Hz rTMS Stimulation — rTMS is an electromagnetic device that provides non-invasive stimulation to the cortex or a sham placebo stimulation that mimics properties without stimulation.
  Other Names: rTMS
Device: Sham rTMS Stimulation — rTMS is an electromagnetic device that provides non-invasive stimulation to the cortex or a sham placebo stimulation that mimics properties without stimulation.

SUMMARY:
This will be a single site pilot study. 30 subjects with Early Phase Psychosis (EPP), defined as medical record documentation of the onset of clinically significant psychotic symptoms within the past ten years, will be enrolled. Prior to randomization (Session 1), subjects will undergo Functional Magnetic Resonance Imaging (fMRI) during Episodic Memory (EM) and Resting State (RS) paradigms. This baseline scan will also include a high-resolution structural sequence for neuronavigation purposes. Then on three separate days each occurring one-week apart, subjects will receive one session of inhibitory (1 Hertz [Hz]) Repetitive Transcranial Magnetic Stimulation (rTMS), one session of excitatory (20 Hz) rTMS, and one sham stimulation session targeting the precuneus. The order of the three interventions will be randomized. Immediately following each rTMS or sham session, subjects will undergo repeat fMRI during EM and RS paradigms. The investigators will also examine the effect of rTMS on EM performance.

DETAILED DESCRIPTION:
In spite of existing work studying rTMS as a treatment modality in schizophrenia, there are no studies that have examined the effects of precuneus directed rTMS on either EM deficits or the neurocircuitry subserving EM in schizophrenia. It is also important to note that the vast majority of studies using rTMS in schizophrenia have examined chronic populations where confounds associated with prolonged duration of illness may be present. Early Phase Psychosis (EPP) is a desirable population to study because these individuals tend to have fewer psychiatric and physical comorbidities and less antipsychotic drug exposure, all of which are factors that may confound investigations of new treatment interventions for this illness. In light of the significant unmet medical need associated with schizophrenia and the grave clinical effect of disrupted EM in the illness, rTMS modulating the precuneus, and potentially EM circuitry, represents an unexplored and potentially novel potential treatment option.

This study proposes to combine functional magnetic resonance imaging (fMRI) with inhibitory Low Frequency (LF) (1 Hz) and excitatory High Frequency (HF) (20 Hz) rTMS protocols to interrogate the effects of rTMS targeting the precuneus on: 1) precuneus activation during EM task performance; 2) functional connectivity between the precuneus and key EM circuitry, specifically the Dorsolateral Prefrontal Cortex (DLPFC), Anterior Cingulate Cortex (ACC), and hippocampus and 3) performance during an in-scanner scene encoding and recognition EM task. This study will provide vital preliminary data on target engagement informing future clinical trials seeking to utilize rTMS to treat EM impairment in schizophrenia. This is an important population for study because if effective, rTMS may represent a novel treatment for EM deficits in schizophrenia. This study will also seek to refine the understanding of the brain circuitry that mediates the potential pro-EM effects of rTMS through the use of fMRI at baseline and following the course of rTMS administration.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 40 years of age
2. Within 10 years of illness onset as defined by entry into treatment for psychotic symptoms
3. Able to give informed consent
4. Willing and able to adhere to the study schedule
5. Structured Clinical Interview for DSM-5 (SCID-5) diagnosis of schizophrenia
6. Clinical stability defined by:

   1. Subjects must not have experienced an exacerbation of their illness within 4 weeks prior to randomization, leading to an intensification of psychiatric care in the opinion of the investigator. Examples of intensification of care include, but are not limited to: inpatient hospitalization, day/partial hospitalization, outpatient crisis management, or psychiatric treatment in an emergency room AND
   2. Antipsychotic treatment stability for at least 4 weeks prior to randomization (no change in antipsychotic dosing or addition of new antipsychotic medication)

Exclusion Criteria:

1. Lifetime history of a seizure, excluding febrile seizures and those induced by substance withdrawal
2. First degree relative with idiopathic epilepsy or other seizure disorder
3. History of significant neurological illness
4. History of head trauma as defined by a loss of consciousness or a post-concussive syndrome
5. Pregnant or breast feeding
6. Known intelligence quotient (IQ) < 70 based on subject report
7. Current acute, serious, or unstable medical conditions
8. Metallic objects planted in or near the head, including implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, Transcutaneous Electrical Nerve Stimulation (TENS) unit, ventriculoperitoneal shunt, or cochlear implants
9. Contraindications to Magnetic Resonance Imaging (MRI) or otherwise unable to tolerate MRI procedures
10. History of electroconvulsive therapy
11. Subjects taking clozapine
12. Subjects who have participated in a clinical trial with any pharmacological treatment intervention for which they received study-related medication in the 4 weeks prior to randomization
13. Subjects considered a high risk for suicidal acts - active suicidal ideation as determined by clinical interview OR any suicide attempt in 90 days prior to screening
14. Current DSM-5 diagnosis of alcohol or drug use disorder (excluding nicotine or caffeine)
15. Subjects who require concomitant treatment with prohibited medication, as specified in Attachment 2

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hummer, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - IU Center for Neuroimaging, Indianapolis, Indiana
  - Prevention and Recovery Center for Early Psychosis, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- rTMS Order 1: 1 Hz rTMS Stimulation First, Then 20 Hz rTMS Stimulation, Then Sham rTMS
- rTMS Order 2: 1 Hz rTMS Stimulation first, then sham rTMS, then 20 Hz rTMS Stimulation
- rTMS Order 3: 20 Hz rTMS Stimulation First, Then 1 Hz rTMS Stimulation, Then Sham rTMS
- rTMS Order 4: 20 Hz rTMS Stimulation First, Then Sham rTMS, Then 1 Hz rTMS Stimulation
- rTMS Order 5: Sham rTMS First, Then 1 Hz rTMS Stimulation, Then 20 Hz rTMS Stimulation
- rTMS Order 6: Sham rTMS first, then 20 Hz rTMS stimulation, then 1 Hz rTMS stimulation
Period: First Intervention (Week 1)
Arm/Group | rTMS Order 1 | rTMS Order 2 | rTMS Order 3 | rTMS Order 4 | rTMS Order 5 | rTMS Order 6
Started | 4 | 5 | 4 | 4 | 3 | 4
Completed | 4 | 5 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (Week 2)
Arm/Group | rTMS Order 1 | rTMS Order 2 | rTMS Order 3 | rTMS Order 4 | rTMS Order 5 | rTMS Order 6
Started | 4 | 5 | 4 | 4 | 3 | 4
Completed | 4 | 5 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (Week 3)
Arm/Group | rTMS Order 1 | rTMS Order 2 | rTMS Order 3 | rTMS Order 4 | rTMS Order 5 | rTMS Order 6
Started | 4 | 5 | 4 | 4 | 3 | 3
Completed | 4 | 5 | 4 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- rTMS Order 1: 1 Hz rTMS stimulation first, then 20 Hz rTMS stimulation, then sham rTMS
  rTMS: Subjects will receive one session of low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of MT, for a total of 1200 pulses.
  Subjects will receive one session of high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minutes.
  Sham: Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
- rTMS Order 2: 1 Hz rTMS stimulation first, then sham rTMS, then 20 Hz rTMS stimulation
  rTMS: Subjects will receive one session of low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of MT, for a total of 1200 pulses.
  Subjects will receive one session of high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minutes.
  Sham: Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
- rTMS Order 3: 20 Hz rTMS stimulation first, then 1 Hz rTMS stimulation, then sham rTMS
  rTMS: Subjects will receive one session of low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of MT, for a total of 1200 pulses.
  Subjects will receive one session of high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minutes.
  Sham: Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
- rTMS Order 4: 20 Hz rTMS stimulation first, then sham rTMS, then 1 Hz rTMS stimulation
  rTMS: Subjects will receive one session of low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of MT, for a total of 1200 pulses.
  Subjects will receive one session of high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minutes.
  Sham: Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
- rTMS Order 5: Sham rTMS first, then 1 Hz rTMS stimulation, then 20 Hz rTMS stimulation
  rTMS: Subjects will receive one session of low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of MT, for a total of 1200 pulses.
  Subjects will receive one session of high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minutes.
  Sham: Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
- rTMS Order 6: Sham rTMS first, then 20 Hz rTMS stimulation, then 1 Hz rTMS stimulation
  rTMS: Subjects will receive one session of low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of MT, for a total of 1200 pulses.
  Subjects will receive one session of high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minutes.
  Sham: Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
- Total: Total of all reporting groups
Arm/Group | rTMS Order 1 | rTMS Order 2 | rTMS Order 3 | rTMS Order 4 | rTMS Order 5 | rTMS Order 6 | Total
Number analyzed (Participants) | 4 | 5 | 4 | 4 | 3 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 4 | 4 | 3 | 4 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (4.08) | 26 (3.08) | 26.5 (4.43) | 23.25 (3.59) | 26 (8.54) | 25.5 (2.38) | 25.21 (4.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 0 | 0 | 1 | 5
  Male | 4 | 4 | 1 | 4 | 3 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 0 | 0 | 1 | 4
  Not Hispanic or Latino | 3 | 4 | 3 | 4 | 3 | 3 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 3 | 2 | 1 | 3 | 13
  White | 3 | 1 | 1 | 2 | 2 | 1 | 10
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 4 | 4 | 3 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Precuneus Functional Activation
Description: Change in estimated beta coefficients for the Target vs. Foil contrast during scene recognition in the precuneus. Beta coefficients reflect the strength of the blood oxygen-level dependent (BOLD) signal during each condition.Target images are those previously shown to participants, and Foil images have not been previously shown, as participants indicate whether they have been shown images. A higher measure indicates that the intervention increased brain activity during recognition of previously shown scenes.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Beta coefficient change (Target vs Foil)
Groups:
- 1 Hz rTMS: Subjects will receive one session of low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of MT, for a total of 1200 pulses.
- 20 Hz rTMS: Subjects will receive one session of high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minutes.
- Sham: Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
Arm/Group | 1 Hz rTMS | 20 Hz rTMS | Sham
Number analyzed (Participants) | 24 | 24 | 23
Beta coefficient change (Target vs Foil) | 0.0329 (0.112) | 0.067 (0.203) | -0.010 (0.112)
Statistical Analysis 1: Comparison: 1 Hz rTMS vs 20 Hz rTMS; Paired t-test comparing Target vs. Foil activity following 1Hz rTMS to Target vs. Foil activity following 20 Hz rTMS stimulation; Test type: Superiority; p = 0.32, t-test, 2 sided — Not adjusted for multiple comparisons; Mean Difference (Net) = -0.042, 95% CI 2-sided [-0.129 to 0.044]
Statistical Analysis 2: Comparison: 1 Hz rTMS vs Sham; Paired t-test between Target vs. Foil activation following 1 Hz rTMS and Target vs. Foil activation following Sham stimulation; Test type: Superiority; p = 0.25, t-test, 2 sided — Not adjusted for multiple comparisons; Mean Difference (Net) = 0.043, 95% CI 2-sided [-0.03 to 0.12]
Statistical Analysis 3: Comparison: 20 Hz rTMS vs Sham; Paired t-test between Target vs. Foil activity following 20 Hz rTMS and Target vs. Foil activity following Sham stimulation; Test type: Superiority; p = 0.13, t-test, 2 sided — Not adjusted for multiple comparisons; Mean Difference (Net) = 0.078, 95% CI 2-sided [-0.024 to 0.181]

2. Primary Outcome: Precuneus Functional Connectivity
Description: Blood oxygen level dependent (BOLD) signal functional connectivity with the precuneus in the bilateral dorsolateral prefrontal cortex, hippocampus, and anterior cingulate cortex. Value is the mean Fisher's transform of the correlation of BOLD time-series in the precuneus with the BOLD time-series in other named regions. Higher values indicate greater connectivity with the precuneus following the intervention. Value of zero indicates no relationship (no connectivity). This value has no unit of measurement.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Transformed correlation coefficient
Groups:
- 1 Hz rTMS: rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of MT, for a total of 1200 pulses.
- 20 Hz rTMS: rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minutes.
Arm/Group | 1 Hz rTMS | 20 Hz rTMS | Sham
Number analyzed (Participants) | 24 | 24 | 23
Transformed correlation coefficient | 0.0657 (0.0394) | 0.0482 (0.0322) | 0.0566 (0.0441)
Statistical Analysis 1: Comparison: 1 Hz rTMS vs 20 Hz rTMS; Paired t-test comparing precuneus connectivity following 1Hz rTMS to precuneus connectivity following 20 Hz rTMS stimulation; Test type: Superiority; p = 0.038, t-test, 2 sided — Not corrected for multiple comparisons; Mean Difference (Net) = 0.018, 95% CI 2-sided [0.001 to 0.034]
Statistical Analysis 2: Comparison: 1 Hz rTMS vs Sham; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Net) = 0.009, 95% CI 2-sided [-0.015 to 0.033]
Statistical Analysis 3: Comparison: 20 Hz rTMS vs Sham; Paired t-test comparing precuneus connectivity following 20Hz rTMS to precuneus connectivity following sham stimulation; Test type: Superiority; p = 0.25, t-test, 2 sided; Mean Difference (Net) = -0.012, 95% CI 2-sided [-0.032 to 0.009]

3. Primary Outcome: Performance During In-scanner Episodic Memory Task
Description: Percent accuracy (0-100%) on detecting whether an image shown during a scene recognition was among those shown during the previous five-minute session. Higher scores indicate better performance in recalling images.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Percentage correct
Arm/Group | 1 Hz rTMS | 20 Hz rTMS | Sham
Number analyzed (Participants) | 24 | 24 | 23
Percentage correct | 80.58 (15.4) | 76.63 (22.4) | 75.61 (20.0)
Statistical Analysis 1: Comparison: 1 Hz rTMS vs 20 Hz rTMS; Paired t-test of scene recognition performance accuracy following 1Hz rTMS to accuracy following 20 Hz rTMS; Test type: Superiority; p = 0.20, t-test, 2 sided — Not adjusted for multiple comparisons; Mean Difference (Net) = 2.7, 95% CI 2-sided [-1.6 to 6.9]
Statistical Analysis 2: Comparison: 1 Hz rTMS vs Sham; Paired t-test of scene recognition performance accuracy following 1Hz rTMS to accuracy following sham rTMS; Test type: Superiority; p = 0.17, t-test, 2 sided — Not corrected for multiple comparisons; Mean Difference (Net) = 4.0, 95% CI 2-sided [-1.9 to 9.9]
Statistical Analysis 3: Comparison: 20 Hz rTMS vs Sham; Paired t-test of scene recognition performance accuracy following 20Hz rTMS to accuracy following 20 Hz rTMS; Test type: Superiority; p = 0.77, t-test, 2 sided — Not adjusted for multiple comparisons; Mean Difference (Net) = -1.3, 95% CI 2-sided [-10.8 to 8.2]

ADVERSE EVENTS:
Time Frame: 1 month
Description: Investigator evaluated for adverse events at every visit
Groups:
- 1 Hz rTMS Stimulation; 20 Hz rTMS Stimulation; Sham rTMS Stimulation: rTMS: Subjects will receive one session of low frequency rTMS within the following stimulation parameters: Continuous 20-minute train of 1 Hz rTMS, at 120% of MT, for a total of 1200 pulses.
  Subjects will receive one session of high frequency rTMS within the following stimulation parameters: 20 Hz, at 120% of MT, 60 trains (1.0 second per train), 20 pulses per train, inter-train interval of 15 seconds, for a total of 1200 pulses over 16 minutes.
  Sham: Sham stimulation session targeting the precuneus. The active and sham functions share the same acoustic properties and sham mimics cutaneous stimulation, facilitating double-blinding.
Arm/Group | 1 Hz rTMS Stimulation | 20 Hz rTMS Stimulation | Sham rTMS Stimulation
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 1/24 | 1/24 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Hz rTMS Stimulation (N=24) | 20 Hz rTMS Stimulation (N=24) | Sham rTMS Stimulation (N=24)
Numbness of fingers (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Application site discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/13/NCT04182113/Prot_SAP_000.pdf